CLINICAL TRIAL: NCT06035510
Title: Effect of Whey Protein Supplementation on Postoperative Outcomes After Gynecological Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 143/2556
Record Dates: First submitted 2023-08-21; First posted 2023-09-13 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2023-08

CONDITIONS: Whey Protein; Postoperative Outcomes; Gynecological Cancer Surgery
Keywords: Whey Protein; Postoperative outcomes; Gynecological Cancer Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- whey protein supplement (Experimental): Participants are given lactose-free Isolated whey protein 23 gm (containing with whey protein isolate 98.7 % ,Soya lecithin 1.3 % ) which mixed with water 350 ml at 6 p.m prior to surgery and 6.00 a.m. at first day after post surgery
  Interventions: Dietary Supplement: whey protein supplement
- standard operative care (No Intervention): Participants followed standard operative care

INTERVENTIONS:
Dietary Supplement: whey protein supplement — Participants are given Isolated whey protein supplement in evening before surgery and first day of post operation to compare with standard operative care on postoperative outcomes after gynecological cancer surgery
  Arms: whey protein supplement

SUMMARY:
Major surgeries including gynecological cancer surgery can make surgical stress that leads to increased burden of postoperative complications, delayed length of hospital stay and increased mortality rate. Protein is one of the essential factors that contribute to the recovery of patients following surgery, as the surgical process increases protein breakdown in the body. Providing patients with an adequate amount of protein helps enhance muscle building, aids in muscle repair, and reduces postoperative inflammation.

One study administered a fluid containing a combination of whey protein and carbohydrates to cancer patients in preoperative and postoperative periods. The result of the study shows that intervention group can reduce the length of hospital stay and postoperative complications.

However, studies focusing on the use of only-protein supplement to improve surgical complications in gynecological cancer patients are limited. This study aims to investigate the administration of protein supplement before and after surgery in gynecological cancer patients its contribution to the reduction of length of hospital stay and postoperative complications at Rajavithi Hospital.

DETAILED DESCRIPTION:
During admission, Participants will be randomized by a computer program into two groups as the whey protein supplement group and control group. Both groups will undergo nutritional assessment on the first day of admission before surgery by the Rajavithi Subjective Global Assessment tool and serum albumin level.

The whey protein supplement group : participants will receive isolated whey protein in the form of two packets of isolated whey protein powder (each packet containing 11.5 grams, totaling to 23 grams) mixed with water in a 350 milliliter drinking bottle at 6.00 p.m. on first day before operation. After the operation, participants will receive the same form of protein supplement as before surgery at 6.00 a.m. on the first day after operation.

The control group : participants will receive standard care, which includes fasting from food after midnight on the night before surgery and other standard surgical protocols.

After surgery, participants will be assessed based on

1. Intraoperative outcomes, which include the duration of surgery, intraoperative blood loss, and intraoperative complications.
2. The postoperative outcomes, which include length of hospital stay, duration of stay in the intensive care unit (ICU), postoperative complications, postoperative pain, time to first ambulation , time to first flatus , nausea and vomiting symptoms, increased requests for pain medication, fever more than 24 hours after surgery , wound infection and readmission.
3. The nutritional status outcomes, assessed through serum albumin levels before surgery and on the 3rd day after surgery in both groups of participants.
4. The side effects of whey protein supplement, in the experimental group participants, which will evaluate include allergic reactions, nausea, vomiting, abdominal discomfort, bloating, headache, reduced appetite, elevated creatinine levels, and increased liver function levels on the 3rd day and two weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. A Woman who suspected or diagnosed with ovarian and endometrial Cancer
2. A Woman who candidates for elective Surgical staging of Laparotomy operation in Rajavithi hospital
3. Aged 18-70 years old
4. Can communicate and understand Thai language very well
5. A woman voluntarily participated in the research

Exclusion Criteria:

1. Allergy to whey protein and protein product such as cow milk and egg
2. A Woman who diagnosed with Hypertension, Diabetes Mellitus, Chronic Kidney Disease, Heart disease and Chronic liver disease
3. A Woman who expected difficult operation such as severe pelvic adhesion or required other surgeon for co-evaluation
4. Pregnant woman or breastfeeding
5. A Woman who denied surgery
6. A Woman who currently take a protein supplement
7. A Woman who take Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) , Bisphosphonates, Levodopa ,Tetracycline and Quinolone

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Length of post-operative hospital stay | an average of 3 days after operation
  Length of post-operative hospital stay after operation to discharged

SECONDARY OUTCOMES:
operative time | start to end of operation, an average of 3 hours
  To compare operative time between intervention group and control group
ICU admission | an average of 3 days after operation
  Length of ICU admission after operation
number of wound infection | 1 and 2 week after operation
  To compare number of wound infection after operation
Readmission | 1 month after operation
  To compare readmission between intervention group and control group
Level of serum albumin | one day before operation and 3 day after operation
  To compare serum albumin before operation and after operation
Side effect of protein supplement | 3 day and 2 week after operation
  To study the side effect of protein supplement
Unit of blood transfusion | start to end of operation, an average of 3 hours
  To compare unit of blood transfusion during operation between intervention group and control group
Intraoperative complication | start to end of operation, an average of 3 hours
  To compare intraoperative complication
postoperative complication | Any events occur within 14 days
  To compare postoperative complication between intervention group and control group
Level of pain score | up to 3 days after operation
  To compare postoperative pain score
time of first ambulation | up to 3 days after operation
  To compare time of first ambulation after operation
time of first flatus and defecation | up to 3 days after operation
  To compare time of first flatus and defecation after operation
Number of additional pain control drug | up to 3 days after operation
  To compare Number of additional pain control drug after operation
Body temperature | Any events occur within 14 days
  To compare post operative fever after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi, Phaya Thai, ratchathewi, Thailand